CLINICAL TRIAL: NCT01508741
Title: Supplement 5-ALA And Sleep And Mood Study
Brief Title: Use Of The Dietary Supplement 5-ALA And Its Relationship With Sleep And Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: SBI ALApromo Co., Ltd. - Strategic Business Innovator (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CHS-19719
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Insomnia; Nocturnal Awakening; Irritability; Coping Behavior; Stress
Keywords: Insomnia; Frequent Nocturnal Awakening; Irritability; Moody; Moodiness; Coping Ability; Coping Behavior; Stress; Feeling Overwhelmed
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-Aminolevulinic Acid (5-ALA) (Active Comparator): Active component 50 mg. capsules of 5-Aminolevulinic Acid (5-ALA)
  Interventions: Dietary Supplement: 5-Aminolevulinic Acid (5-ALA)
- Placebo capsule (Placebo Comparator): Non-active component capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 5-Aminolevulinic Acid (5-ALA) — 5-ALA 50 mg. p.o. daily capsules taken over 6 weeks.
  Other Names: 5-Aminolevulinic Acid; 5-ALA
  Arms: 5-Aminolevulinic Acid (5-ALA)
Dietary Supplement: Placebo — Daily p.o. capsule of similar shape and color to active ingredient 5-ALA capsule taken over 6 weeks.
  Arms: Placebo capsule

SUMMARY:
PURPOSE: The purpose of this investigation is to determine if a relationship exists between the administration of a dietary supplement containing 5-ALA and sleep and mood.

HYPOTHESIS: There are several possible mechanisms for improvement in sleep and mood. In one study involving test mice, researchers found that the regular administration of 5-ALA appeared to raise serotonin levels in the brain. One hypothesis is by increasing serotonin levels, 5-ALA may contribute to improvements with sleep, along with additional improvements in mood, calmness, irritability and coping abilities. 5-ALA may also support hormonal regulation, including melatonin, in the pineal gland and corticosteroid regulation in the adrenal glands.

Another hypothesis is that 5-ALA may have an impact on increasing the energy and metabolism of cells, such that its own circadian rhythms are better defined. 5-ALA may support neuronal function and assistance with "mental energy" needed to deal with stress in daily life, producing better feelings of "coping", "less irritability" and lowering an individual's feelings of "fatigue", all of which may contribute to a reduction of "pessimism" regarding the ability to deal with daily tasks.

DESIGN: This will be a double-blinded, randomized parallel-group comparison study.

SAMPLE: 40 participants will be randomized to the following 2 study groups for each outcome variable (Sleep and Mood): Control Group - 20 participants and Intervention Group - 20 participants. A table of random numbers will be used to assign the participants.

DETAILED DESCRIPTION:
5-Aminolevulinic Acid (5-ALA) is a dietary supplement and a naturally occurring amino acid. It is a natural delta amino acid; as a non-alpha amino acid, it is not a component of proteins. 5-ALA is synthesized in the mitochondria, and is the first compound in the prophyrin synthesis pathway, the pathway that leads to heme in mammals and chlorophyll in plants. 5-ALA has been associated with genetic information, structure and metabolism, and energy conversion.

5-ALA can be found in many common foods, such as spinach, tomatoes, shitake mushrooms, potatoes, squid, ground beef, wine and soy sauce. The normal intake from food containing 5-ALA is 1-2 mg/day. 5-ALA is synthesized by the body at a rate of 600 mg/day.

Data has supported the hypothesis that supplementation with 5-ALA may be related to improved sleep, mood and coping abilities. This research study will further explore this potential relationship.

The duration of the study for each participant is a total of 10 weeks, which include 4 separate appointments, spaced 3-4 weeks apart. Participants in the Intervention Group will begin taking one daily 50 mg capsule p.o. of 5-ALA over a 6 week period, and the Control Group will be provided with a placebo of similar size and color.

Before entering the research study, each participant undergoes a thorough screening process, including lab work (CBC and Ferritin). Once accepted into the study, the daily capsules are started and a diary is filled out by each participant at home each day and brought to each appointment for review. Instructions are given to record patterns and changes pertaining to sleep, mood or coping abilities. After 6 weeks, the participant is then instructed to stop the daily capsules but to continue daily diary recordings. They are also scheduled for one final appointment at week 10. At each of the 4 appointments over the 10 week period, assessments are performed by health care professionals, questionnaires and daily diaries are reviewed/recorded and anthropometric measurements are obtained.

The product used in this investigation contains 3 components:

* 5-Aminolevulinic acid (5-ALA) phosphate
* Sodium Ferrous Citrate (SFC)
* Corn starch as filler.

The 5-ALA capsules and contents are Non-GMO, BSE free, and alcohol free. The products tested are manufactured under food GMP conditions. A certificate of analysis is available.

Variables monitored as part of the evaluation will be assessed by comparing the intervention group to the control group. Two-sample t-tests will be used to assess statistical significance at baseline and follow-up exams. Baseline data will be summarized as means and standard deviations with differences among the randomized groups tested for significance by t-tests and chi-square tests. To measure the possible differences in rates of change in sleep and mood scores across follow-up time between the 5-ALA treatment and the control group, additional analyses will estimate differences in slopes using linear regression models. Mixed linear models will be fit using the proc mixed procedure in SAS 9.2. The regression models will include an indicator variable identifying treatment groups, a variable for weeks of follow-up, and interaction terms between the indicator variables and follow-up time. Results will be summarized as the difference in slopes comparing the intervention groups to the control group. Results will also be presented graphically to illustrate the estimated differences in slopes for the study groups. All significant tests will be two-sided.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults Living On Oahu, Hawaii (or able to personally attend five/1-hour/on-site appointments on Oahu, over a 10 week period)
* No Medication Or Supplements Currently Taken For Sleep Or Mood Adjustments
* Body Weight 110-250 Pounds
* Normal CBC And Ferritin Labwork Done At Screening
* All Participants Self-Reporting Insomnia, Nocturnal Awakening, Difficulty Sleeping/Falling Asleep Or Feeling Moody

Exclusion Criteria:

* Participants With A History Of Hepatitis, Porphyria, Hemochromatosis, Or Iron Sensitivity
* Participants With Active Liver Disease
* Women Who Are Pregnant Or Breastfeeding
* Participants Currently In Another Clinical Study
* Labwork With Ferritin Levels Elevated Above 125% Of Normal On Screening

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
5-ALA Supplementation And Its Relationship To Sleep And Mood | 10 weeks
  Patterns relating to sleep and mood will be recorded each day of the study by each participant over a 10 week period. This study is conducted to determine if a daily 50 mg p.o. intake of 5-ALA reveals a relationship of improvement regarding patterns of sleep or mood.

CONTACTS AND LOCATIONS:
Overall Officials: Rosanne C. Harrigan, Ed.D., Study Chair — University of Hawaii at Manoa, John A. Burns School of Medicine, Dept. of Complementary and Alternative Medicine; Beatriz L. Rodriguez, M.D., Principal Investigator — University of Hawaii at Manoa, John A. Burns School of Medicine, Dept. of Complementary and Alternative Medicine and Dept. of Geriatric Medicine; Terry Shintani, M.D., Study Director — University of Hawaii at Manoa, John A. Burns School of Medicine, Dept. of Complementary and Alternative Medicine
Locations (1):
- University of Hawaii at Manoa, John A. Burns School of Medicine, Dept. of Complementary and Alternative Medicine, Honolulu, Hawaii, United States